CLINICAL TRIAL: NCT06485453
Title: Predictive Urodynamic Parameters for The Treatment Efficacy of Onabotulinum A Toxin in Neurogenic Lower Urinary Tract Dysfunction
Status: Completed | Type: Observational
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Muharrem Baturu, Assistant Proffesor, University of Gaziantep
Other Study IDs: GAUN-Urology-Baturu-001
Record Dates: First submitted 2024-06-25; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Neurogenic Bladder Disorder
Keywords: Onabotulinumtoxin A; Neurogenic lower urinary tract dysfunction; Urodynamics
MeSH Terms: conditions — Urinary Bladder, Neurogenic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Botulinum Toxin A responder: Patients who respond to the 200 IU Onabotulinum toxin-A injections were allocated to Groups 1
  Interventions: Drug: Botox 200 UNT Injection
- Botulinum Toxin A non-responder: Patients who did not respond to the 200 IU Onabotulinum toxin-A injections were allocated to Groups 2
  Interventions: Drug: Botox 200 UNT Injection

INTERVENTIONS:
Drug: Botox 200 UNT Injection — Treatment effect and duration of Onabotulinum Toxin A according to patient's pad usaged

SUMMARY:
Purpose: To evaluate urodynamic parameters predicting the treatment efficacy of onabotulinumtoxin A (onaBoNT-A) in patients with neurogenic lower urinary tract dysfunction (NLUTD).

Methods: Patients with NLUTD who received 200 IU onaBont-A injections at Gaziantep University, Faculty of Medicine, Department of Urology between September 2013 and September 2023 were included in the study. Urodynamic parameters, including cystometric capacity, detrusor pressure (Pdet), and compliance, detrusor leak point pressure (DLPP), phasic or terminal neurogenic overactivity were assessed. Additionally, the correlations between these parameters and treatment outcomes were analyzed.

Changes in the number of pads used per day due to UI were assessed every 3 months during the postoperative period. The time lapsed to return to the pad usage levels before onaBoNT-A injections was recorded as the duration of the benefit.

Preoperative urodynamic data of the patients were compared between groups. Additionally, a subgroup analysis was conducted in patients who benefited from treatment to evaluate the correlation between treatment efficacy, duration of benefit from treatment, and urodynamic parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Neurogenic Lower Urinary Tract Disorder
* Aged >18 years
* Patients who did not respond adequatel to antimuscarinics or could not tolerate their side effects
* Antimuscarinic treatment failure with at least two different antimuscarinic agents for a minimum of 3 months.

Exclusion Criteria:

* Patients with Lower Urinary Tract Disorder due to functional or non-neurogenic etiologies
* Patients who received onaBoNT-A doses either other than 200 IU or its multiple doses
* In the 12-month period designated for patient follow-up, patients who did not attend their check-ups

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Neurogenic Lower Urinary Tract Disorder who didn't respond to anticholinergic treatment were the goal population.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Number of patients after onabotulinum a toxin injections who respond to treatment | received 200 IU of onaBoNT-A injections for the first time, and followed up regularly for the duration of at least 12 months.

SECONDARY OUTCOMES:
treatment succes duration of patients | Received 200 IU of onaBoNT-A injections for the first time, and followed up regularly for the duration of at least 12 months.
  The duration of the decrease in the number of pads used was calculated

IPD SHARING:
Plan to Share IPD: No